CLINICAL TRIAL: NCT01974180
Title: Smoking-induced EGF-dependent Reprogramming of Airway Basal Cell Function
Status: Terminated | Type: Observational
Why Stopped: Closed by investigator
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1305013972; Weill Cornell Medical College (Other Grant/Funding Number: Weill Cornell Medical College)
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Smoking; COPD; Chronic Obstructive Pulmonary Disease
Keywords: Smoking; COPD; Chronic Obstructive Pulmonary Disease; Healthy Smoker; Non-smoker
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Airway epithelial samples collected under IRB protocol #1204012331 will be used.
Oversight: Data Monitoring Committee: No

SUMMARY:
Early changes associated with the development of smoking-induced diseases, e.g., COPD and lung cancer (the two commonest causes of death in U.S.) are often characterized by abnormal airway epithelial differentiation. Airway basal cells (BC) are stem/progenitor cells necessary for generation of differentiated airway epithelium. Based on our preliminary observations that epidermal growth factor receptor, known to regulate airway epithelial differentiation, is enriched in BC and its ligand EGF is induced by smoking, we hypothesized that smoking-induced EGF alters the ability of BC to form normally differentiated airway epithelium. To test this, airway BC will be purified using a cell-culture method established in our laboratory and responses to EGF will be analyzed using genome-wide microarrays and an in vitro air-liquid interface model of airway epithelial differentiation.

DETAILED DESCRIPTION:
Airway epithelium is composed of 4 major cell types, including ciliated cells, secretory cells, undifferentiated columnar cells, and basal cells (BC). The earliest changes associated with the development of smoking-induced lung diseases, such as chronic obstructive pulmonary disease (COPD) and lung cancer, occur in the airway epithelium, including BC hyperplasia, squamous metaplasia, mucous cell hyperplasia and metaplasia, impaired ciliated cell structure and function, loss of Clara cells, and increased epithelial permeability due to impaired junctional barrier. We hypothesize that fundamental to these changes are smoking-induced derangements of BC, the stem/progenitor cell population that can self-renew and differentiate into ciliated and secretory cells. Using technologies established in our laboratory to culture pure population of BC from the human airway epithelium, to induce differentiation of these BC in air-liquid interface, and to assess the transcriptome of purified BC compared to that of the complete differentiated airway epithelium, our preliminary data indicates that: (1) airway BC exhibit a distinct gene expression signature relevant to stem/progenitor cell function, including high expression of the epidermal growth factor receptor (EGFR); (2) airway BC from healthy smokers have a different gene expression pattern compared to nonsmokers, with enrichment of functional categories related to cell cycle and proliferation and down-regulation of differentiation-associated genes; and (3) constitutive EGF expression in BC and differentiated cells is barely detectable, but smoking selectively up-regulates EGF expression in differentiated cells of the airway epithelium in vivo. Based on these data and on the knowledge that EGFR signaling plays a central role in the regulation of cell proliferation and differentiation in the airway epithelium, the central concept of this proposal is that smoking-induced expression by differentiated cells activates BC via EGFR altering the molecular phenotype of airway BC and impairing their ability to generate normal differentiated airway epithelium. To assess this concept, the following aims will be addressed:

Aim 1. To determine whether stimulation of airway BC from healthy nonsmokers with EGF induces genes and pathways related to smoking-associated phenotypes, e.g. BC hyperplasia, squamous metaplasia, mucous metaplasia, abnormal cilia, decreased Clara cell number and compromised junctional integrity.

Aim 2. To test the hypothesis that stimulation of airway BC from healthy nonsmokers with EGF alters BC differentiation in air-liquid interface culture, with generation of smoking-associated phenotypes (see Aim 1).

Aim 3. To test the hypothesis that upon apical exposure to cigarette smoke extract, differentiated airway epithelial cells derived from BC of healthy nonsmokers release increased amounts of EGF into the apical supernatant, which will alter the ability of BC of healthy nonsmokers to generate normal differentiated airway epithelium, and that blocking EGF in this supernatant will abolish this effect.

ELIGIBILITY:
Inclusion Criteria:

* Must be capable of providing informed consent
* Males and females, age 18 or older
* Good overall health without history of chronic lung disease, including asthma, and without recurrent or recent (within 3 months) acute pulmonary disease
* Normal physical examination
* Normal routine laboratory evaluation, including general hematologic studies, general serologic/ immunologic studies, general biochemical analyses, and urine analysis
* Negative HIV serology
* Normal chest X-ray (PA and lateral)
* Normal electrocardiogram
* Females - not pregnant
* No history of allergies to medications to be used in the bronchoscopy procedure
* Not taking any medications relevant to lung disease or having an effect on the airway epithelium Willingness to participate in the study

Exclusion Criteria:

* Unable to meet the inclusion criteria
* Pregnancy
* Current active infection or acute illness of any kind
* Current alcohol or drug abuse
* Evidence of malignancy within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-23 (Actual)

PRIMARY OUTCOMES:
EGF induced gene expression changes related to smoking-associated phenotypes | One year
  To determine whether stimulation of airway BC from healthy nonsmokers with EGF induces genes and pathways related to smoking-associated phenotypes, e.g. BC hyperplasia, squamous metaplasia, mucous metaplasia, abnormal cilia, decreased Clara cell number and compromised junctional integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Renat Shaykhiev, MD, PHD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided